CLINICAL TRIAL: NCT05193955
Title: The Effect of Laughter Yoga Practiced Before Simulation Training on State Anxiety, Student Satisfaction and Perceived Stress Level of Undergraduate Nursing Students
Brief Title: The Effect of Laughter Yoga Practiced Before Simulation Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe ARIKAN DÖNMEZ, Asst. Prof., Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: KA-20027
Record Dates: First submitted 2021-11-26; First posted 2022-01-18 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Laughter; State Anxiety; Stress; Self Confidence; Satisfaction, Personal
MeSH Terms: conditions — Laughter; Anxiety Disorders; Personal Satisfaction | interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): undergraduate students who practice laughter yoga and simulation education together
  Interventions: Other: Laughter Yoga
- Control Group (No Intervention): undergraduate students who practice simulation education

INTERVENTIONS:
Other: Laughter Yoga — Laughter yoga is one of the methods that is among the complementary therapy and supportive care practices in the world and is used increasingly. Laughter yoga is a non-invasive and non-pharmacological method that combines unconditional laughter with yoga breathing techniques. In laughter yoga, one can laugh without being humorous, joking, or funny. Laughter is simulated by starting out as a physical exercise and making eye contact with other members of the group and playing games with them. The body cannot distinguish between real and unreal laughter and laughter begins.
  Arms: Intervention Group

SUMMARY:
Simulation education has become one of the innovative educational approaches that are widely used in providing nursing students with knowledge, skills, and attitudes towards vocational courses. Simulation education provides students with the opportunity to combine their knowledge and skills and provide nursing care in a high-reality environment. However, the fact that simulation training is a method that requires the student to recognize a clinical event, make a clinical decision, and intervene with the patient in line with this decision may cause students to experience anxiety and affect their learning. Although there are limited studies conducted on nursing students, it is stated that new approaches such as laughter yoga are effective in reducing anxiety and stress levels. In this direction, this research; In this study, it was planned to investigate the effectiveness of laughter yoga in terms of reducing the anxiety experienced by nursing students during simulation training and increasing their learning satisfaction. The universe of the research will be the second-year students of Hacettepe University Faculty of Nursing. As a result of the power analysis, it is aimed to reach 54 people. The study was planned in a randomized controlled design. Research data will be collected through Personal Information Form, State Anxiety Scale, Student Satisfaction and Self-Confidence in Learning Scale, Perceived Stress Scale for Nursing Students, and Students' Vital Findings Evaluation Form. With this study, it is predicted that laughter yoga to be applied to nursing students before simulation training will have a positive effect on state anxiety, student satisfaction, and perceived stress level.

DETAILED DESCRIPTION:
The study will be carried out in a randomized controlled design with the aim of determining the effect of laughter yoga applied before the simulation training on the state anxiety, student satisfaction, and perceived stress level of nursing students. After the power analysis to calculate the sample size of the study, a total of 36 students will be included in each group with 90% power and 5% margin of error for multiple variance analysis in repeated measurements in a 2x2 factorial pattern between groups. In the research, students who have applied laughter yoga and simulation application together will form the intervention group, and students who only participated in the simulation application will form the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Students who voluntarily agree to participate in the research will be included in the research.

Exclusion Criteria:

* Taking any medication that affects the heart rate,
* Having any psychiatric disease such as anxiety disorder,
* Students who do not accept to participate in the research will not be included in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
State Anxiety Scale | It will be applied to the students just before simulation and/or laughter yoga and after completing the training on the same day (each session is 60 minutes). Change from baseline State Anxiety scores at the end of 60 minutes.
  Inventory is used to determine how an individual feels at a particular moment and in a situation.High scores indicate high anxiety level, low scores indicate low anxiety level. There are two types of statements in the scale, direct and reverse. Direct statements express negative emotions, reversed statements express positive emotions. Reversed statements are items 1,2,5,8,10,11,15,16,19 and 20. After finding the total weights of the direct and reversed statements separately, a predetermined and unchanging value (50) is added to the result obtained by subtracting the total weight score of the reverse statements from the total weight score obtained for the direct statements.Range of scores for each subtest is 20-80, the higher score indicating greater anxiety.

SECONDARY OUTCOMES:
Student Satisfaction and Self-Confidence in Learning Scale | It will be applied immediately after completing the simulation training and/or laughter yoga on the same day (at the end of 60 minutes). Change from baseline Student Satisfaction and Self-Confidence in Learning scores at the end of 60 minutes.
  This scale, which is widely used to evaluate students' attitudes and beliefs about simulation, was published by the National League for Nurses. The Turkish validity-reliability study of the scale was carried out by Karaçay and Kaya in 2017. Accordingly, the Cronbach's Alpha coefficient of the scale was found to be 0.88. There are two sub-dimensions, "satisfaction with learning" and "self-confidence", and a total of 13 items in the scale. The highest total score that can be obtained from the scale is 65, and the lowest is 13.The high score that can be obtained from the total of the scale indicates high satisfaction and self-confidence.
Perceived Stress Scale for Nursing Students | It will be applied to the students just before simulation and/or laughter yoga and after completing the training on the same day (each session is 60 minutes). Change from baseline Perceived Stress scores at the end of 60 minutes.
  The Perceived Stress Scale for Nursing Students (PSASS), a 29-item scale originally in Chinese, was developed by Sheu et al. It was developed by (2002) . The Turkish validity-reliability study of the scale was performed by Karaca et al. (2015) made by Accordingly, the Cronbach's Alpha coefficient of the scale was found to be 0.85. The total score that can be obtained from the scale ranges from 0 to 116. As the score obtained from the scale increases; perceived stress level also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe ARIKAN DÖNMEZ, PhD, Principal Investigator — Hacettepe University Faculty of Nursing
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No